CLINICAL TRIAL: NCT02743637
Title: A Phase 1 Dose Escalation Study of SDX-7320 to Assess the Safety and Tolerability in Patients With Advanced Refractory or Late-Stage Solid Tumors
Brief Title: A Dose Escalation Study of SDX-7320 in Patients With Advanced Refractory or Late-Stage Solid Tumors
Acronym: SDX-0101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SynDevRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDX-0101
Record Dates: First submitted 2016-04-07; First posted 2016-04-19 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Advanced Malignancy; Advanced Solid Tumors; Neoplasm; Metastasis
Keywords: Cancer; Oncology; Solid Tumors; Phase 1; SDX-7320; SynDevRx; MetAP2; Breast; Post menopausal; Colorectal; Pancreatic; Ovarian; Endometrial; Esophageal; Lung; Renal; Prostate; Liver
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SDX-7320 (Experimental): Increasing dose cohorts, until the maximum tolerated dose (MTD) is determined.
  Interventions: Drug: SDX-7320

INTERVENTIONS:
Drug: SDX-7320 — SDX-7320 is a synthetic copolymer-drug conjugate of a novel MetAP2 inhibitor.

SUMMARY:
This is a Phase 1 dose escalation to assess the safety, tolerability and maximum tolerated dose of subcutaneous administered SDX-7320 in patients with advanced refractory or late-stage solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1 dose escalation study to assess the safety and tolerability of subcutaneously administered SDX-7320 in patients with advanced refractory or late-stage solid tumors.

Once the MTD has been determined up to 12 patients will be treated at this dose level, to further characterize treatment emergent adverse events (TEAEs).

ELIGIBILITY:
Inclusion Criteria:

* Patients have at least one site of radiographically measurable disease.
* Eastern Cooperative Oncology Group (ECOG) status ≤1.
* Adequate renal and liver functions.
* Life expectancy ≥3 months.

Exclusion Criteria:

* Patients that have undergone organ transplant surgery.
* The patient has a known history of Hepatitis A, B, or C and is on active anti-viral therapy.
* History of gastric bypass surgery or banding procedure.
* Uncontrolled or refractory hypertension: systolic >180 or diastolic >110, or hypotension: systolic <90 or diastolic <50 despite medical treatment.
* Participation in any other trial of an investigational agent within 30 days prior to first dose of study drug.
* The resting 12-lead electrocardiogram obtained during screening shows QTc (Fridericia correction) ≥470 ms or has a congenital prolonged QT syndrome.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of SDX-7320 to find the recommended Phase II dose | Up to 30 days after last subject enrolled

SECONDARY OUTCOMES:
Anti-tumor activity | From the screening visit though the end of the last cycle on treatment, an expected average of 16 weeks
  RECIST v1.1

OTHER OUTCOMES:
Peak plasma concentration (Cmax) of active moiety SDX7539 | Cycle 1, 3, and 6 Day 1: predose, 3, 6, 24, 48, 96 hours; Cycle 2, 4, and 5: predose
Area under the plasma concentration curve from zero to infinity AUC (0-inf) active moiety SDX7539 | Cycle 1, 3, and 6 Day 1: predose, 3, 6, 24, 48, 96 hours; Cycle 2, 4, and 5: predose

CONTACTS AND LOCATIONS:
Overall Officials: Neal Salomon, MD, Study Director — SynDevRx, Inc.
Locations (3):
- United States (3):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Sponsor Website — http://syndevrx.com